CLINICAL TRIAL: NCT01862328
Title: A Phase 1b, Open-Label, Dose Escalation, Multi-arm Study of MLN4924 Plus Docetaxel, Gemcitabine, or Combination of Carboplatin and Paclitaxel in Patients With Solid Tumors
Brief Title: Dose Escalation, Multi-arm Study of MLN4924 Plus Docetaxel, Gemcitabine, or Combination of Carboplatin and Paclitaxel in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C15010; U1111-1220-1470 (Other: WHO)
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumors
Keywords: MLN4924; Solid Tumors
MeSH Terms: interventions — pevonedistat; Paclitaxel; Gemcitabine; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MLN4924 and Docetaxel (Arm 1) (Experimental)
  Interventions: Drug: MLN4924; Drug: Docetaxel
- MLN4924 + Paclitaxel + Carboplatin (Arm 2) (Experimental)
  Interventions: Drug: MLN4924; Drug: Paclitaxel; Drug: Carboplatin
- MLN4924 + Gemcitabine (Arm 3) (Experimental)
  Interventions: Drug: MLN4924; Drug: Gemcitabine

INTERVENTIONS:
Drug: MLN4924 — MLN4924 (intravenously [IV]) in participants in a 21-day cycle:
  * MLN4924 on Days 1,3,5 of each cycle
  Other Names: Pevonedistat
Drug: Paclitaxel — Paclitaxel (IV) in a 21-day cycle:
  * Paclitaxel on Day 1 of each cycle
  Arms: MLN4924 + Paclitaxel + Carboplatin (Arm 2)
Drug: Gemcitabine — Gemcitabine (IV) in participants in a 28-day cycle:
  -Gemcitabine on Days 1,8,15 of each cycle
  Arms: MLN4924 + Gemcitabine (Arm 3)
Drug: Docetaxel — Docetaxel (IV) in participants in a 21-day cycle:
  - Docetaxel on Day 1 of each cycle
  Arms: MLN4924 and Docetaxel (Arm 1)
Drug: Carboplatin — Carboplatin (IV) in participants in a 21-day cycle:
  - Carboplatin on Day 1 of each cycle
  Arms: MLN4924 + Paclitaxel + Carboplatin (Arm 2)

SUMMARY:
The purpose of this study is to establish the maximum tolerated dose (MTD) and assess the safety and tolerability of MLN4924 (pevonedistat) in combination with docetaxel, paclitaxel and carboplatin, and gemcitabine in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
3. Have a histologically or cytologically confirmed metastatic or locally advanced and incurable solid tumor that is felt to be appropriate for treatment with 1 of the 3 chemotherapy regimens in this study, or have progressed despite standard therapy, or for whom conventional therapy is not considered effective. The tumor must be radiographically or clinically evaluable and/or measurable
4. Recovered (that is, <=Grade 1 toxicity) from the effects of prior antineoplastic therapy
5. Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to practice true abstinence
6. Male participants who agree to practice effective barrier contraception or agree to practice true abstinence
7. Voluntary written consent must be given before performance of any study-related procedure
8. Suitable venous access for the study-required blood sampling
9. Adequate clinical laboratory values during the screening period as specified in the protocol
10. Participants who are willing to refrain from donating blood for at least 90 days after their final dose of MLN4924 and (for male participants) willing to refrain from donating semen for at least 4 months after their final dose of MLN4924
11. Availability of fixed tumor specimen (block or slides) for exploratory biomarker analysis. If no slides or block are available, fresh tumor biopsies should be obtained and used for these assessments

Exclusion Criteria:

1. Major surgery within 14 days before the first dose of study drug
2. Female participants who are lactating or pregnant
3. Active uncontrolled infection or severe infectious disease
4. Receiving antibiotic therapy within 14 days before the first dose of study treatment
5. Life-threatening illness unrelated to cancer
6. Known hypersensitivity to study-assigned chemotherapy
7. Prior treatment with MLN4924; however, prior treatment with docetaxel, paclitaxel,carboplatin, and gemcitabine is allowed
8. History of severe hypersensitivity reactions to docetaxel (polysorbate 80-based formulations) for participants to be enrolled in Arm 1 (MLN4924 + docetaxel), history of hypersensitivity to carboplatin for participants to be enrolled in Arm 2 (MLN4924 + paclitaxel + carboplatin), or history of severe hypersensitivity to paclitaxel (cremophor-based formulations) for participants to be enrolled in Arm 2
9. Persistent diarrhea (greater than Grade 2) lasting >3 days within 2 weeks before the first dose of study treatment
10. Systemic antineoplastic therapy within 21 days before the first dose of study drug
11. Radiotherapy within 14 days preceding the first dose of study treatment
12. Prior treatment with radiation therapy involving greater than or equal to (>=) 25% of the hematopoietically active bone marrow
13. Treatment with cytochrome P450 3A (CYP3A) inducers within 14 days before the first dose of MLN4924.

Treatment with CYP3A inhibitors within 14 days before the first dose of MLN4924; however, voriconazole and fluconazole need only be stopped for 3 days before MLN4924. Participants must have no history of amiodarone use in the 6 months before the first dose of MLN4924 14. Clinically uncontrolled central nervous system (CNS) involvement 15. Any serious medical or psychiatric illness 16. Treatment with any investigational products 21 days prior to treatment 17. Unwilling or unable to refrain from using statins 24 hours before, the day of, and 24 hours after each MLN4924 administration 18. Known human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection 19. Known hepatic cirrhosis 20. Known cardiac/cardiopulmonary disease 21. Left ventricular ejection fraction 23. with a cardiac pacer whose heart rate is set at a fixed rate and participants on concomitant medication that may limit increase in heart rate in response to hypotension 24 History of severe intolerance to cytotoxic agent(s) given in the assigned arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Atlanta, Georgia
  - St Louis, Missouri
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Faessel HM, Mould DR, Zhou X, Faller DV, Sedarati F, Venkatakrishnan K. Population pharmacokinetics of pevonedistat alone or in combination with standard of care in patients with solid tumours or haematological malignancies. Br J Clin Pharmacol. 2019 Nov;85(11):2568-2579. doi: 10.1111/bcp.14078. Epub 2019 Sep 4. PMID 31355467
- [Derived] Lockhart AC, Bauer TM, Aggarwal C, Lee CB, Harvey RD, Cohen RB, Sedarati F, Nip TK, Faessel H, Dash AB, Dezube BJ, Faller DV, Dowlati A. Phase Ib study of pevonedistat, a NEDD8-activating enzyme inhibitor, in combination with docetaxel, carboplatin and paclitaxel, or gemcitabine, in patients with advanced solid tumors. Invest New Drugs. 2019 Feb;37(1):87-97. doi: 10.1007/s10637-018-0610-0. Epub 2018 May 21. PMID 29781056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 10 June 2013 to 21 May 2018.
Pre-assignment Details: Participants with solid tumors were enrolled to receive MLN4924 in combination with docetaxel (Arm 1), paclitaxel + carboplatin (Arm 2), or gemcitabine (Arm 3) during the Dose-escalation and maximum tolerated dose (MTD) expansion portion of this study. Participants in Lead-in cohort received MLN4924 + carboplatin only (Arm 2a).
Groups:
- Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2: MLN4924 15 milligram per square meter (mg/m^2), infusion, intravenously, once on Days 1, 3, and 5 and docetaxel 75 mg/m^2, infusion, intravenously, once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or progressive disease (PD) (up to Cycle 52).
- Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2: MLN4924 25 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 and docetaxel 75 mg/m^2, infusion, intravenously, once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
- Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6: MLN4924 15 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 and carboplatin AUC6, infusion intravenously once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
- Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5: MLN4924 15 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 and paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 followed by carboplatin AUC5, infusion, intravenously once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
- Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5: MLN4924 20 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 and paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 followed by carboplatin AUC5, infusion, intravenously once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
- Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5: MLN4924 25 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 and paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 followed by carboplatin AUC5 infusion, intravenously once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
- Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2: MLN4924 25 mg/m^2, infusion, intravenously, once on Days 1, 8, and 15 and gemcitabine 1000 mg/m^2, infusion, intravenously, once on Days 1, 8, and 15 before administration of MLN4924 in a 28-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
Period: Overall Study
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Started | 4 | 18 | 6 | 7 | 12 | 7 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 18 | 6 | 7 | 12 | 7 | 10
Not completed — Progressive Disease | 3 | 11 | 5 | 6 | 7 | 4 | 3
Not completed — Adverse Event | 0 | 4 | 0 | 1 | 0 | 2 | 4
Not completed — Other | 0 | 2 | 1 | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants who received at least 1 dose of any study drug.
Groups:
- Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2: MLN4924 15 milligram per square meter (mg/m^2), infusion, intravenously, once on Days 1, 3, and 5 and docetaxel 75 mg/m^2, infusion, intravenously, once on Day 1 before administration of MLN4924 in a 21-day cycle up to symptomatic deterioration or PD (up to Cycle 52).
- Total: Total of all reporting groups
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2 | Total
Number analyzed (Participants) | 4 | 18 | 6 | 7 | 12 | 7 | 10 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (2.99) | 60.0 (9.82) | 56.8 (9.56) | 58.1 (10.65) | 57.9 (14.34) | 59.0 (12.00) | 59.7 (14.45) | 58.8 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 4 | 4 | 8 | 1 | 4 | 34
  Male | 2 | 7 | 2 | 3 | 4 | 6 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 3 | 14 | 6 | 7 | 11 | 7 | 7 | 55
  Unknown or Not Reported | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 2 | 2 | 1 | 0 | 1 | 12
  White | 3 | 13 | 4 | 5 | 11 | 7 | 9 | 52
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 18 | 6 | 7 | 12 | 7 | 10 | 64
Body surface area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] | 1.9 (0.32) | 1.9 (0.28) | 1.8 (0.29) | 2.0 (0.28) | 1.9 (0.32) | 1.9 (0.17) | 1.9 (0.25) | 1.9 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least 1 Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 5 years)
Population: The safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 4 | 18 | 6 | 7 | 12 | 7 | 10
Participants
  TEAE | 4 | 18 | 6 | 7 | 12 | 7 | 10
  SAE | 1 | 9 | 3 | 2 | 3 | 1 | 7

2. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Laboratory Evaluation Findings
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 5 years)
Population: The safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 4 | 18 | 6 | 7 | 12 | 7 | 10
Participants
  Anaemia | 1 | 4 | 2 | 2 | 7 | 2 | 3
  Aspartate aminotransferase increased | 0 | 6 | 2 | 2 | 5 | 2 | 2
  Alanine aminotransferase increased | 0 | 7 | 1 | 1 | 4 | 1 | 3
  Neutrophil count decreased | 1 | 5 | 1 | 3 | 3 | 1 | 1
  Neutropenia | 1 | 1 | 1 | 1 | 4 | 4 | 3
  Thrombocytopenia | 0 | 1 | 3 | 1 | 3 | 3 | 3
  Platelet count decreased | 0 | 1 | 2 | 3 | 2 | 2 | 3
  White blood cell count decreased | 1 | 2 | 0 | 0 | 4 | 0 | 0
  Hypomagnesaemia | 0 | 2 | 2 | 0 | 0 | 1 | 0
  Blood creatinine increased | 1 | 2 | 0 | 0 | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 2 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 1 | 0 | 0 | 1 | 1 | 0
  Blood bilirubin increased | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Hypophosphataemia | 0 | 2 | 0 | 0 | 1 | 0 | 0
  Hypokalaemia | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Blood glucose increased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Liver function test abnormal | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Haematocrit decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Red blood cell count decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycaemia | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Hyponatraemia | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Vital Sign Findings
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 5 years)
Population: The safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 4 | 18 | 6 | 7 | 12 | 7 | 10
Participants
  Tachycardia | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Hypotension | 1 | 3 | 2 | 2 | 0 | 2 | 1

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: complete disappearance of all target lesions and non-target disease, with exception of nodal disease; all nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 millimeter [mm]); no new lesions. PR: greater than or equal to (>=) 30 percent (%) decrease under baseline of sum of diameters of all target lesions; short axis was used in sum for target nodes, while longest diameter was used in sum for all other target lesions; no unequivocal progression of non-target disease; no new lesions.
Time Frame: Screening, Cycle 2 Days 15 (Arm 1, 2a, and 2) and 22 (Arm 3) then every other Cycle thereafter up to 30 days after the last dose of study drug (up to 5 years) (Cycle Length = 21 days [Arm 1, 2a, and 2] and 28 days [Arm 3])
Population: The response-evaluable population was defined as all the participants who received at least 1 dose of MLN4924, had measurable disease at baseline, and had at least 1 post baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 3 | 16 | 6 | 7 | 11 | 5 | 6
percentage of participants
  CR | 0 | 0 | 0 | 0 | 18 | 0 | 0
  PR | 0 | 19 | 17 | 0 | 36 | 40 | 0

5. Secondary Outcome: Duration of Response
Description: Duration of response: time from the date of first documented response per the investigator response assessment (CR or PR) to the date of PD or the date of last disease assessment if the participant discontinued the study before PD using RECIST 1.1 CR: complete disappearance of all target lesions and non-target disease, with exception of nodal disease; all nodes, both target and non-target, must decrease to normal (short axis <10 mm); no new lesions. PR: >=30% decrease under baseline of sum of diameters of all target lesions; short axis was used in sum for target nodes, while longest diameter was used in sum for all other target lesions; no unequivocal progression of non-target disease; no new lesions. PD: at least a 20% increase (including an absolute increase of at least 5 mm) in sum of diameters of target lesions, taking as reference smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From the date of first documented response (CR or PR) to the date of first documented PD or the date of last disease assessment if the participants discontinued the study before PD (up to 5 years)
Population: The response-evaluable population is defined as all participants who receive at least 1 dose of study drug, have measurable disease at baseline, and have at least 1 post baseline disease assessment. The number of participants analyzed includes only those participants who had data available for this measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 0 | 3 | 1 | 0 | 6 | 2 | 0
months |  | 2.880 (2.7644) | 2.270 (NA) — Standard deviation could not be calculated since only one participant was available for analysis. |  | 16.153 (15.9867) | 7.015 (1.1384) |

6. Secondary Outcome: Dose-escalation Phase: Plasma Concentrations-time Data of MLN4924
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 20 hours) post-dose (Cycle Length=21 days [Arm 1 and 2] and 28 days [Arm 3])
Population: The safety population was defined as all participants who received at least 1 dose of any study drug. The number of participants analyzed includes only those participants who had data available for this measure. This outcome measure was planned to be assessed only in the Dose-escalation phases of Arms 1, 2, and 3.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
Number analyzed (Participants) | 4 | 18 | 7 | 12 | 7 | 10
nanogram per milliliter (ng/ml)
  Cycle 1 Day 1: End-dose: number analyzed (Participants) | 4 | 12 | 7 | 6 | 7 | 10
  Cycle 1 Day 1: End-dose | 163.8 (109.15) | 197.1 (51.94) | 275.7 (98.67) | 257.3 (110.05) | 372.7 (120.93) | 222.0 (87.62)
  Cycle 1 Day 1: 1.5 hours post dose: number analyzed (Participants) | 4 | 12 | 7 | 6 | 7 | 10
  Cycle 1 Day 1: 1.5 hours post dose | 82.0 (39.97) | 130.6 (46.94) | 156.8 (53.46) | 192.7 (80.35) | 246.7 (47.24) | 160.5 (122.07)
  Cycle 1 Day 1: 3 hours post dose: number analyzed (Participants) | 4 | 12 | 7 | 5 | 7 | 10
  Cycle 1 Day 1: 3 hours post dose | 48.0 (12.05) | 95.8 (19.70) | 152.4 (56.19) | 138.0 (73.10) | 186.9 (32.30) | 103.0 (39.00)
  Cycle 1 Day 1: 20 hours post dose: number analyzed (Participants) | 4 | 12 | 7 | 6 | 7 | 10
  Cycle 1 Day 1: 20 hours post dose | 7.5 (1.50) | 14.6 (4.81) | 23.4 (9.19) | 34.6 (25.09) | 24.4 (10.81) | 14.2 (5.09)

7. Secondary Outcome: MTD Expansion Phase: Plasma Concentrations-time Data of MLN4924
Description: The number of participants analyzed includes only those participants who had data available for this measure.
Time Frame: Cycle 1 Days 1 and 5 pre-dose and at multiple time points (up to 20 hours) post-dose (Cycle Length=21 days [Arm 1 and 2])
Population: The safety population was defined as all participants who received at least 1 dose of any study drug. This outcome measure was planned to be assessed for participants who received the MTD in Arms 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5
Number analyzed (Participants) | 18 | 12
ng/ml
  Cycle 1 Day 1: End-dose: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 1: End-dose | 152.8 (83.67) | 429.8 (95.87)
  Cycle 1 Day 1: 1.5 hours post dose: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 1: 1.5 hours post dose | 137.3 (37.19) | 253.6 (19.65)
  Cycle 1 Day 1: 3 hours post dose: number analyzed (Participants) | 6 | 4
  Cycle 1 Day 1: 3 hours post dose | 86.4 (29.16) | 192.8 (39.14)
  Cycle 1 Day 1: 6 hours post dose: number analyzed (Participants) | 0 | 4
  Cycle 1 Day 1: 6 hours post dose |  | 136.3 (14.73)
  Cycle 1 Day 1: 7 hours post dose: number analyzed (Participants) | 6 | 0
  Cycle 1 Day 1: 7 hours post dose | 63.4 (24.87) |
  Cycle 1 Day 1: 20 hours post dose: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 1: 20 hours post dose | 14.2 (5.39) | 30.2 (7.98)
  Cycle 1 Day 5: End-dose: number analyzed (Participants) | 5 | 5
  Cycle 1 Day 5: End-dose | 211.1 (116.43) | 253.2 (56.60)
  Cycle 1 Day 5: 1.5 hours post dose: number analyzed (Participants) | 5 | 4
  Cycle 1 Day 5: 1.5 hours post dose | 115.3 (42.54) | 171.0 (19.44)
  Cycle 1 Day 5: 3 hours post dose: number analyzed (Participants) | 5 | 5
  Cycle 1 Day 5: 3 hours post dose | 96.7 (53.48) | 118.4 (19.69)
  Cycle 1 Day 5: 6 hours post dose: number analyzed (Participants) | 0 | 5
  Cycle 1 Day 5: 6 hours post dose |  | 76.5 (4.97)
  Cycle 1 Day 5: 7 hours post dose: number analyzed (Participants) | 4 | 0
  Cycle 1 Day 5: 7 hours post dose | 38.3 (17.84) |
  Cycle 1 Day 5: 20 hours post dose: number analyzed (Participants) | 4 | 5
  Cycle 1 Day 5: 20 hours post dose | 9.8 (2.07) | 10.9 (3.40)

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug and no more than 30 days (up to 5 years) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/4 | 2/18 | 0/6 | 0/7 | 0/12 | 1/7 | 3/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 9/18 | 3/6 | 2/7 | 3/12 | 1/7 | 7/10
Other Adverse Events (participants affected / at risk) | 4/4 | 18/18 | 6/6 | 6/7 | 12/12 | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 (N=4) | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 (N=18) | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 (N=6) | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 (N=7) | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 (N=12) | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 (N=7) | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2 (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MLN4924 15 mg/m^2 + Docetaxel 75 mg/m^2 (N=4) | Arm 1: MLN4924 25 mg/m^2 + Docetaxel 75 mg/m^2 (N=18) | Arm 2a: MLN4924 15 mg/m^2 + Carboplatin AUC6 (N=6) | Arm 2: MLN4924 15 mg/m^2+Paclitaxel 175mg/m^2+Carboplatin AUC5 (N=7) | Arm 2:MLN4924 20 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 (N=12) | Arm 2:MLN4924 25 mg/m^2+Paclitaxel 175 mg/m^2+Carboplatin AUC5 (N=7) | Arm 3: MLN4924 25 mg/m^2 + Gemcitabine 1000 mg/m^2 (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 6 | 3 | 2 | 8 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 1 | 3 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 4 | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 8 | 5 | 3 | 8 | 3 | 5
Constipation (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 5 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 1 | 4 | 6 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1 | 3 | 6 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 2 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 11 | 4 | 5 | 7 | 5 | 4
Pyrexia (General disorders) | 1 | 4 | 1 | 1 | 2 | 3 | 2
Oedema peripheral (General disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 3
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 3 | 2 | 1
Pain (General disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 4 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 2 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 2 | 2 | 5 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 7 | 1 | 1 | 4 | 1 | 4
Neutrophil count decreased (Investigations) | 1 | 4 | 1 | 3 | 3 | 1 | 1
Platelet count decreased (Investigations) | 0 | 1 | 2 | 3 | 2 | 2 | 3
White blood cell count decreased (Investigations) | 1 | 2 | 0 | 0 | 5 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 4 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 0 | 0 | 2 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 3 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0 | 3 | 3 | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 2 | 2 | 1 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 1 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0 | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 3 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2 | 6 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 1 | 3 | 4 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 2 | 4 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 0 | 1 | 5 | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 2 | 3 | 0 | 2 | 2 | 1
Headache (Nervous system disorders) | 0 | 3 | 2 | 0 | 2 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 3 | 2 | 1 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 2 | 1 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 3 | 5 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 3 | 2 | 3 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 2 | 2 | 0 | 2 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular appendage torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT01862328/SAP_000.pdf
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT01862328/Prot_001.pdf